CLINICAL TRIAL: NCT07202260
Title: Pragmatic Analysis of Complex Radiotherapy Cases In Cancer of the Lung (The PRACTICAL Study)
Brief Title: Pragmatic Analysis of Complex Radiotherapy Cases In Cancer of the Lung
Acronym: PRACTICAL
Status: Active, not recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSP 230
Record Dates: First submitted 2025-02-20; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (NSCLC); Lung Cancer (SCLC)
Keywords: radiotherapy; interstitial lung disease; vascular invasion; re-irradiation; rare histology
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with co-existing interstitial lung disease
- Patients who undergo radiotherapy twice to the same area (reirradiation).
- Patients with the less common or rare types of lung cancer
- Patients with cancer invading large blood vessels.
- Patients with oligopersistent/oligoprogressive disease on immunotherapy or targeted therapies.

SUMMARY:
This study focuses on improving care for people with lung cancer who face unusual or complex treatment situations.

DETAILED DESCRIPTION:
By studying detailed patient data, researchers aim to find the best ways to treat these patients while reducing short- and long-term side effects. The findings will help refine radiotherapy treatments, ensuring they are as safe and effective as possible. Additionally, the results will provide doctors with better information to help patients understand the potential risks and benefits of their treatment options.

ELIGIBILITY:
Inclusion Criteria: Complex patients with lung cancer undergoing radiotherapy in one of the following groups;

* Rare histology
* Disease invading vascular structures
* Co-existing interstitial lung disease (ILD)
* Radical re-irradiation
* Oligopersistent/oligoprogressive disease on immunotherapy or targeted therapies.

Exclusion Criteria:

* Include patients with stage IV disease who are receiving non-curative intent radiotherapy
* There are no exclusion criteria relating to upper age limit or comorbidities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, with stage I, II or III lung cancer undergoing curative-intent radiotherapy at the Christie Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute and late toxicity | 2 years
  - Acute (<90 days post radiotherapy) and late (> 90 days post radiotherapy) toxicity according to common terminology criteria for adverse events (CTCAE) V5.

OTHER OUTCOMES:
Patient reported quality of life | 2 years
  - Patient reported quality of life (QOL) information from electronic patient reported outcome measure (ePROM) questionnaires.
Survival | 2 years
  - Progression-free survival and overall survival.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Withington, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No